CLINICAL TRIAL: NCT07259603
Title: Association Between Vitamin D Deficiency and Disease Activity in Patients With Inflammatory Bowel Disease
Brief Title: Association Between Vitamin D Deficiency and Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hamed Gadelrab, principal investigator, Assiut University
Other Study IDs: ADIBD
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with Crohn's disease (CD) and ulcerative colitis (UC): Adults aged ≥18 years, diagnosed with Crohn's disease (CD) and ulcerative colitis (UC), and on regular follow-up in the IBD clinic, are followed up for recent vitamin D and disease activity assessment (within 1 month)
  Interventions: Diagnostic Test: Serum 25(OH)D (Vitamin D3), C- reactive protein, Erthrocyte sedimentation rate

INTERVENTIONS:
Diagnostic Test: Serum 25(OH)D (Vitamin D3), C- reactive protein, Erthrocyte sedimentation rate — Serum 25(OH)D (Vitamin D3), C- reactive protein, Erthrocyte sedimentation rate are evaluated to assess vitamin D deficiency and IBD activity

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are two major types of inflammatory bowel disease (IBD) that are identified by different clinical, endoscopic, pathological, and radiologic diagnostic methods.

In the past few years, the incidence of inflammatory bowel disease has been increasing worldwide, with the incidence of UC being higher than that of CD.

Vitamin D is a fat-soluble vitamin that is produced in the skin by a UV-dependent reactionand then hydroxylated by the kidneys and liver, and is converted to its active form, 1,25-dihydroxyvitamin D.

Vitamin D deficiency is common throughout the world and its deficiency rates ranging from 30 to 50% have been reported.

Several studies have shown the role of vitamin D as a regulator of the immune system and its inhibitory function incellular immunity and production of pro-inflammatory cytokines that play a major role in autoimmune diseases.

In some human studies, the link between vitamin D levels and the disease severity of IBD has been shown, but it is not clear whether lack of vitamin D is the cause or consequence.

In this study, we aimed to investigate the relationship between inflammatory bowel disease and itsflare-up with serum levels of vitamin D

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Diagnosed with crohn's and ulcerative colitis
* Regular follow-up in IBD clinic
* Recent vitamin D and disease activity assessment (within 1 month)

Exclusion Criteria:

* Current vitamin D supplementation(>1000IU/day)

  * History of malabsorption syndromes (e.g.,celiac disease)
  * Chronic kidney or liver disease
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adults aged ≥18 years
  * Diagnosed with crohn's and ulcerative colitis
  * Regular follow-up as an outpatient in the IBD clinic at Al-RAGHI hospital Assuit university
  * Recent vitamin D and disease activity assessment (within 1 month)
  * Sample Size Calculation:
  Assuming an expected prevalence of vitamin D deficiency in IBD patients around 50%, a sample size of n = 100-150 will give adequate power (80%) to detect significant correlations (p < 0.05) between vitamin D levels and disease activity indices.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of vitamin D deficiency in patients with active inflammatory bowel disease | Recent vitamin D and disease activity assessment (within 1 month)
  This will be done by measuring the vitamin D level in the serum of patients with active inflammatory bowel diseases (in nanograms/ milliliter)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Cantorna MT, Zhu Y, Froicu M, Wittke A. Vitamin D status, 1,25-dihydroxyvitamin D3, and the immune system. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1717S-20S. doi: 10.1093/ajcn/80.6.1717S. PMID 15585793
- [Background] Cantorna MT. Vitamin D and its role in immunology: multiple sclerosis, and inflammatory bowel disease. Prog Biophys Mol Biol. 2006 Sep;92(1):60-4. doi: 10.1016/j.pbiomolbio.2006.02.020. Epub 2006 Feb 28. PMID 16563470
- [Background] Mouli VP, Ananthakrishnan AN. Review article: vitamin D and inflammatory bowel diseases. Aliment Pharmacol Ther. 2014 Jan;39(2):125-36. doi: 10.1111/apt.12553. Epub 2013 Nov 17. PMID 24236989
- [Background] Fletcher J, Cooper SC, Ghosh S, Hewison M. The Role of Vitamin D in Inflammatory Bowel Disease: Mechanism to Management. Nutrients. 2019 May 7;11(5):1019. doi: 10.3390/nu11051019. PMID 31067701